CLINICAL TRIAL: NCT06834269
Title: Efficacy of Transcranial Static Magnetic Field Stimulation (tSMS) and Potential Theranostic Biomarkers in Amyotrophic Lateral Sclerosis (ALS).
Brief Title: Transcranial Static Magnetic Stimulation (tSMS) and Potential Theranostic Biomarkers in Amyotrophic Lateral Sclerosis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Di Lazzaro Vincenzo, Full Professor of Neurology, Campus Bio-Medico University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StaticALS
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyothrophic Lateral Sclerosis; ALS; tSMS; transcranial magnetic stimulation; NF-L; YKL-40; p75ECD; Biomarkers; transcranial static magnetic stimulation; TDP43
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pwALS (Experimental): All participants will undergo tSMS administration at home, in two daily sessions of 120 minutes each.
  Interventions: Device: Transcranial magnetic stimulation (tSMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (tSMS) — Transcranial static magnetic stimulation (tSMS) will be delivered simultaneously to both hemispheres, at the motor cortex (M1), via magnets housed in a helmet.

SUMMARY:
The objective of the present study is to assess the efficacy of tSMS in ALS patients. This will be achieved by monitoring:

* levels of NF-L and other potential innovative biomarkers,
* clinical progression, trough ALSFRS-R. After at least three-month follow-up, participants will be recruited to undergo biemispheric tSMS for two daily sessions of 120 minutes each, at home, for 12 months. Together with clinical status, which will be evalueted each three months, blood and urine samples will be collected before the start of the tSMS administration (M0) and during the treatment (M3, M6, M9, M12), to detect potential theranostic biomarkers. In a subgroup of patients, ad additional blood and urine sample will be collected 3 months before M0 (M-3).

Moreover, cortical excitability will be tested through transcranial magnetic stimulation (TMS) before and after the tSMS stimulation period.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* diagnosis of possible, probable or definite ALS according to revised El Escorial criteria and Awaji-Shima criteria
* disease duration < 24 months
* ALSFRS-R > 30 at the recruitment
* ALSFRS-R decline > 1 in the at least 3-months period before the intervention
* normal respiratory functionality at the preliminary evaluation (M-3), assessed in the previous month (FVC ≥ 75% and ALSFRS-R items 10,11,12 > 4)
* treatment with riluzole 50 mg x 2/die

Exclusion Criteria:

* inclusion in other clinical trials
* presence of tracheotomy or/and PEG (percutaneous endoscopic gastrostomy)
* unable to perform spirometry due to severe bulbar involvement
* contraindications to magnetic fields exposure
* pregnancy or breastfeeding
* history of epilepsy or seizures
* use of drugs acting on central nervous system, except for antidepressive drugs and benzodiazepines.
* cognitive impairment
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
NfL reduction | 12 months
  The potential reduction of NfL during treatment is monitored by blood samples collected at baseline, and then , every 3 months during the treatment

SECONDARY OUTCOMES:
Monthly Progression Rate (MPR) | 15 months
  MPR is derived from the comparison between the ALSFRS-R (Revised Amyotrophic Lateral Sclerosis Functional Rating Scale) decline over the period of at least three months before the treatment, and the period of twelve months during the treatment. The ALSFRS-R is 12-items scale ranking from 0 (worse) to 48 (better) points.
New Potential Theranostic Biomarkers Assay | 12 months
  Investigation of potential theranostic biomarkers in blood samples (YKL-40, TDP43) and urine samples (p75ECD), collected at baseline and evrey three months during the treatment
Effect on resting motor threshold (RMT) and active motor threshold (AMT) | 12 months
  Change in TMS-derived cortical excitability parameters (RMT and AMT) before and after stimulation period.
Effect on motor evoked potentials (MEP) size | 12 months
  Change in TMS-derived cortical excitability parameters (MEP size) before and after stimulation period.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Campus Bio-Medico, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided